CLINICAL TRIAL: NCT01018472
Title: Probiotics in Infants With Cyanotic Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 200917427
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Cyanotic Congenital Heart Disease
Keywords: cyanotic heart disease; congenital heart disease; intestinal microbiota; probiotics
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bifidobacterium infantis (Experimental)
  Interventions: Dietary Supplement: Bifidobacterium infantis
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Bifidobacterium infantis — 1 billion organisms twice daily either through a feeding tube or by mouth for 4 months
  Arms: Bifidobacterium infantis
Other: Placebo — A dilute preparation of pregestimil formula (similar in appearance to the probiotic product)
  Arms: Placebo

SUMMARY:
Infants with congenital heart disease have more frequent infections and exposures to antibiotics than healthy infants. It is unknown how congenital heart disease affects the development of bacterial colonization of the intestines. It is also unknown whether probiotics will change the bacteria in the intestine of infants with heart disease to become more like those of healthy infants without heart disease. This pilot trial is designed to address these two questions.

DETAILED DESCRIPTION:
Infants with cyanotic congenital heart disease will be randomly assigned to receive either a placebo or probiotic Bifidobacterium infantis. Comparisons will be made between the infants receiving the placebo and healthy infants without heart disease and between the infants receiving the placebo and those receiving the probiotic.

ELIGIBILITY:
Inclusion Criteria:

* Cyanotic congenital heart disease
* Term infant
* Born at or transferred to UC Davis Children's hospital

Exclusion Criteria:

* Congenital anomalies of the intestinal tract

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2009-11; Primary Completion 2011-02 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Fecal microbiota | Weekly for 4 weeks then monthly

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Underwood, MD, Principal Investigator — UC Davis School of Medicine
Locations (1):
- UC Davis Children's Hospital, Sacramento, California, United States